CLINICAL TRIAL: NCT05196568
Title: Pilot Study on the Effects of Fasting Mimicking Diet (FMD) in Women With Polycystic
Brief Title: Effects of Fasting Mimicking Diet (FMD) in Women With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Salento (Other)
Responsible Party: Principal Investigator, Anna Maria Giudetti, Principal Investigator, University of Salento
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VERBALE N° 56
Record Dates: First submitted 2021-12-07; First posted 2022-01-19 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-01

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients not treated with the mimic fasting diet (No Intervention): Group treated with the mimic fasting diet
- patients treated with the mimic fasting diet (Experimental): Group treated with the mimic fasting diet
  Interventions: Dietary Supplement: Fasting mimicking diet

INTERVENTIONS:
Dietary Supplement: Fasting mimicking diet — Women will be given three administrations of fasting mimicking diet once a month
  Arms: patients treated with the mimic fasting diet

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy in reproductive-aged women, affecting 6-21% (depending on the applied diagnostic criteria) of this population worldwide. PCOS is characterized by hyperandrogenism and/or chronic anovulation which can manifest with a range of symptoms (e.g., hirsutism, acne, oligomenorrhea, and infertility) and is associated with increased risk of cardiometabolic diseases, including hypertension, dyslipidemia, insulin resistance (IR), and type 2 diabetes mellitus (T2DM). Moreover, PCOS is linked to increased psychological morbidity (e.g., increased risk of stress, depression, low self-esteem, and poor body image). The exact PCOS etiology is unknown, but increased adiposity is considered pivotal. Indeed, almost 90% of women with PCOS are overweight or obese, and even moderate weight loss may result in clinically meaningful improvements in hyperandrogenism and menstrual regularity. Also, women with PCOS often have more severe IR than weight-matched women without PCOS, whilst their increased susceptibility to obesity may further exacerbate IR and the accompanying metabolic and reproductive dysfunctions. As such, women with PCOS exhibit an increased risk of impaired glucose tolerance and T2DM regardless of weight and age. Management of overweight/obese women with PCOS focuses on weight loss through regular exercise and diet, aiming to alleviate its clinical manifestations and lower the related risk of T2DM and cardiovascular disease. Fasting-induced negative energy also potently affects the hormones such as estradiol, testosterone, and leptin, and complex interactions exist between metabolic signals and ovarian steroids. However, fasting is difficult to implement. It is of great interest to develop feasible and efficacious fasting-mimicking diets (FMD) to alleviate the burden of fasting while preserving the beneficial effects of fasting. In a case study, the investigators observed that a 23-year-old female diagnosed with PCOS had her persistent cystic acne resolved after just 3 cycles of self-administered fasting-mimicking dieting. In addition, FDM induces a reduction in insulin levels, fasting glucose, BMI, decreased adiposity, and inflammation rates. The investigators hypothesize that a specially designed FMD will induce physiological changes similar to prolonged fasting and will decrease risk factors associated with metabolic syndrome and alleviate symptoms of PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy in reproductive-aged women, affecting 6-21% (depending on the applied diagnostic criteria) of this population worldwide. PCOS is characterized by hyperandrogenism and/or chronic anovulation which can manifest with a range of symptoms (e.g., hirsutism, acne, oligomenorrhea, and infertility) and is associated with increased risk of cardiometabolic diseases, including hypertension, dyslipidemia, insulin resistance (IR), and type 2 diabetes mellitus (T2DM). Moreover, PCOS is linked to increased psychological morbidity (e.g., increased risk of stress, depression, low self-esteem, poor body image, and reduced health-related quality of life). The exact PCOS etiology is unknown, but increased adiposity is considered pivotal. Indeed, almost 90% of women with PCOS are overweight or obese, and even moderate weight loss (e.g., 5%) may result in clinically meaningful improvements in hyperandrogenism and menstrual regularity. Also, women with PCOS often have more severe IR than weight-matched women without PCOS, whilst their increased susceptibility to obesity may further exacerbate IR and the accompanying metabolic and reproductive dysfunctions. As such, women with PCOS exhibit an increased risk of impaired glucose tolerance and T2DM regardless of weight and age. Management of overweight/obese women with PCOS focuses on weight loss through regular exercise and diet, aiming to alleviate its clinical manifestations and lower the related risk of T2DM and cardiovascular disease. Fasting-induced negative energy also potently affects the hormones such as estradiol, testosterone, and leptin; and complex interactions exist between metabolic signals and ovarian steroids. However, fasting is difficult to implement. It is of great interest to develop feasible and efficacious fasting-mimicking diets (FMD) to alleviate the burden of fasting while preserving the beneficial effects of fasting. In a case study, a 23-year-old female diagnosed with PCOS had her persistent cystic acne resolved after just 3 cycles of self-administered fasting-mimicking dieting. In addition, FDM induces a reduction in insulin levels, fasting glucose, BMI, decreased adiposity, and inflammation rates. The investigators hypothesize that a specially designed FMD will induce physiological changes similar to prolonged fasting and will decrease risk factors associated with metabolic syndrome and alleviate symptoms of PCOS.

The purpose of the study is to evaluate the effect of FMD in women with PCOS. Regarding the study model, a crossover will be applied. Our crossover design is the simplest model known as 2 x 2 where two treatments are compared in two-period, two-sequence model. Each washout, between consecutive periods, is done so that the previous treatment does not affect the response to the next treatment. The main advantage of a crossover design over the parallel group is the opportunity it offers to compare the effects of treatments within-subjects, which is not possible with a conventional parallel-group design. Additionally, a crossover design usually requires a smaller sample size to reliably estimate the magnitude of the treatment effect. That is, any component of an individual's response that is consistent over time is removed from the treatment comparison. Study participants will be randomized and assigned to arm 1 (n° = 50, control patients) or arm 2 (n° = 50, patients undergoing FMD). Patients in the FMD group will be asked to consume FMD, which will be provided with a box, for 5 continuous days, and to return to their normal diet after completion until the next cycle which will start 25 days later, for a total of three months.

The two groups will then be exchanged in the third month so that the control group will also be subjected to FMD in the following three months.

The main parameters that will be texted, are all major symptoms associated with PCOS, including menstrual cycle regularity, ovarian morphology (by ultrasound); hirsutism (by the Ferriman-Gallwey (FG) scoring method), and acne score. Moreover, improvement in metabolic, inflammatory, and psychological markers will be also evaluated.

Both control and FMD patients will complete anthropometric measurements every month (at the end of each FMD cycle). After three months, patients will be crossed for another 3 months: patients with arm 1 control will be instructed to follow FMD, while patients with arm 2 undergoing FMD will be asked to continue their normal diet. Follow-up exams will be conducted for both groups at the end of the 6th month. Thereafter, all patients will be asked to continue their normal diet for another three months and will undergo further follow-up at the end of the ninth month. Blood chemistry analyzes will be performed at time zero, at 3 and 6 months, while gynecological and nutritional checks will be performed at time zero at 3 to 6 months and at the end of the study (t = 9 months). The total duration of the study is 9 months. The evaluation of the menstrual history and the anthropometric parameters will be measured during the gynecological and nutritional checks. The psychological/psychiatric evaluation will be carried out at T0, at 3 to 6 months, and at 9 months. Blood samples will also be used for IGF-1 analyzes (IFOM, Milan). Both control and FMD patients will fill out a food diary. Patients undergoing FMD will be contacted by phone for nutritional assistance once a day during the 5 days of FMD. Additionally, to assess adherence to the 5-day nutritional plan for FMD, patients will independently assess their ketonuria with appropriate sticks. Every month, all enrolled patients will note the possible date of menstruation and the duration of the cycle.

ELIGIBILITY:
Inclusion Criteria:

* Female 18-40 years
* BMI 20-40
* Reproductive age women with PCOS diagnosis
* Irregular menstrual cycles

  * Chronic oligo/anovulation defined as an intermenstrual interval of >45 days
  * < 8 menstrual cycles/year
  * evidence of either hyperandrogenemia (elevation of total or free testosterone above the normal range for women)
  * clinical hyerandrogenism (hirsutism and or acne)
* 3 years from menarche
* Agree to avoidance of pregnancy and to use barrier contraception for duration of study

Exclusion Criteria:

* • Clinically ascertained presence of type I and type II Diabetes

  * Pregnancy and/or nursing
  * Medication exclusion

    * Use of medications and/or supplements that influence either ovarian function or insulin sensitivity, within 2 months: including oral contraceptive pills, hormonal implants, anti-androgens, antipsychotics or antihypertensives metformin, glucocorticoids, and/or health food remedies other than multi-vitamins and calcium;
    * Subjects who are on oral contraception, metformin, or nutritional supplements must agree to discontinue these drugs and undergo an 8 week washout period before the tests are performed
    * Other drugs that cannot be suspended during the FMD phase
  * Alcohol usage more than 7 drinks/week

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Restoration of menstrual regularity | End of the treatment (three months)
  The main parameter that will be taken into consideration as an improvement of the syndrome is the restoration of the menstrual cycle, which is not regular in the woman with polycystic ovary syndrome

SECONDARY OUTCOMES:
Improvement of blood glucose values (mg / dl) | End of the treatment (three months)
  All improvements in glycemia values that are generally increased in polycystic ovary syndrome are considered
Improvement of blood insulinemic values (µU/mL) | End of the treatment (three months)
  Improvements in the parameter that is generally increased in polycystic ovary
Improvement of blood glycated hemoglobin (%) | End of the treatment (three months)
  Improvements in the parameter that is generally increased in polycystic ovary
Improvement of blood LDL, HDL, total cholesterol and triglycerides (mg/dl) | End of the treatment (three months)
  All improvements in plasma lipid parameters that are generally modified in polycystic ovary
Improvement in plasma sexual hormones | End of the treatment (three months)
  Improvements in plasma values of FSH, LH, E2, SHBG, Total Testosterone, DHEA-S, Δ4androstenedione, TSH, generally altered in polycystic ovary
Improvemet in the PCR value | End of the treatment (three months)
  Improvements in inflammatory parameters that are modified in polycystic ovary syndrome are considered
Improvement in depression syntoms evaluated bu Basic Self- Esteem Scale and improvement in quality of life, assessed by WHOQOL-BREF test | End of the treatment (three months)
  Improvements of the parameters related to the psychiatric sphere that are modified in the polycystic ovary syndrome are considered

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Giudetti, Principal Investigator — University of Salento
Locations (1):
- Anna Maria Giudetti, Lecce, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azziz R, Carmina E, Chen Z, Dunaif A, Laven JS, Legro RS, Lizneva D, Natterson-Horowtiz B, Teede HJ, Yildiz BO. Polycystic ovary syndrome. Nat Rev Dis Primers. 2016 Aug 11;2:16057. doi: 10.1038/nrdp.2016.57. PMID 27510637
- [Background] Balen AH, Conway GS, Kaltsas G, Techatrasak K, Manning PJ, West C, Jacobs HS. Polycystic ovary syndrome: the spectrum of the disorder in 1741 patients. Hum Reprod. 1995 Aug;10(8):2107-11. doi: 10.1093/oxfordjournals.humrep.a136243. PMID 8567849
- [Background] Boyle JA, Cunningham J, O'Dea K, Dunbar T, Norman RJ. Prevalence of polycystic ovary syndrome in a sample of Indigenous women in Darwin, Australia. Med J Aust. 2012 Jan 16;196(1):62-6. doi: 10.5694/mja11.10553. PMID 22256938
- [Background] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889
- [Background] Costello M, Shrestha B, Eden J, Sjoblom P, Johnson N. Insulin-sensitising drugs versus the combined oral contraceptive pill for hirsutism, acne and risk of diabetes, cardiovascular disease, and endometrial cancer in polycystic ovary syndrome. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD005552. doi: 10.1002/14651858.CD005552.pub2. PMID 17253562
- [Background] Dunaif A, Segal KR, Futterweit W, Dobrjansky A. Profound peripheral insulin resistance, independent of obesity, in polycystic ovary syndrome. Diabetes. 1989 Sep;38(9):1165-74. doi: 10.2337/diab.38.9.1165. PMID 2670645
- [Background] Ehrmann DA, Liljenquist DR, Kasza K, Azziz R, Legro RS, Ghazzi MN; PCOS/Troglitazone Study Group. Prevalence and predictors of the metabolic syndrome in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2006 Jan;91(1):48-53. doi: 10.1210/jc.2005-1329. Epub 2005 Oct 25. PMID 16249284
- [Background] Glueck CJ, Dharashivkar S, Wang P, Zhu B, Gartside PS, Tracy T, Sieve L. Obesity and extreme obesity, manifest by ages 20-24 years, continuing through 32-41 years in women, should alert physicians to the diagnostic likelihood of polycystic ovary syndrome as a reversible underlying endocrinopathy. Eur J Obstet Gynecol Reprod Biol. 2005 Oct 1;122(2):206-12. doi: 10.1016/j.ejogrb.2005.03.010. PMID 16219521
- [Background] Himelein MJ, Thatcher SS. Depression and body image among women with polycystic ovary syndrome. J Health Psychol. 2006 Jul;11(4):613-25. doi: 10.1177/1359105306065021. PMID 16769740
- [Background] Holte J, Bergh T, Berne C, Wide L, Lithell H. Restored insulin sensitivity but persistently increased early insulin secretion after weight loss in obese women with polycystic ovary syndrome. J Clin Endocrinol Metab. 1995 Sep;80(9):2586-93. doi: 10.1210/jcem.80.9.7673399.
- [Background] Kiddy DS, Sharp PS, White DM, Scanlon MF, Mason HD, Bray CS, Polson DW, Reed MJ, Franks S. Differences in clinical and endocrine features between obese and non-obese subjects with polycystic ovary syndrome: an analysis of 263 consecutive cases. Clin Endocrinol (Oxf). 1990 Feb;32(2):213-20. doi: 10.1111/j.1365-2265.1990.tb00857.x. PMID 2112067
- [Background] Kumar S, Kaur G. Intermittent fasting dietary restriction regimen negatively influences reproduction in young rats: a study of hypothalamo-hypophysial-gonadal axis. PLoS One. 2013;8(1):e52416. doi: 10.1371/journal.pone.0052416. Epub 2013 Jan 29. PMID 23382817
- [Background] Legro RS, Kunselman AR, Dodson WC, Dunaif A. Prevalence and predictors of risk for type 2 diabetes mellitus and impaired glucose tolerance in polycystic ovary syndrome: a prospective, controlled study in 254 affected women. J Clin Endocrinol Metab. 1999 Jan;84(1):165-9. doi: 10.1210/jcem.84.1.5393. PMID 9920077
- [Background] Legro RS, Kunselman AR, Dunaif A. Prevalence and predictors of dyslipidemia in women with polycystic ovary syndrome. Am J Med. 2001 Dec 1;111(8):607-13. doi: 10.1016/s0002-9343(01)00948-2. PMID 11755503
- [Background] Ma YM, Li R, Qiao J, Zhang XW, Wang SY, Zhang QF, Li L, Tu BB, Zhang X. Characteristics of abnormal menstrual cycle and polycystic ovary syndrome in community and hospital populations. Chin Med J (Engl). 2010 Aug;123(16):2185-9. PMID 20819662
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] Norman RJ, Masters L, Milner CR, Wang JX, Davies MJ. Relative risk of conversion from normoglycaemia to impaired glucose tolerance or non-insulin dependent diabetes mellitus in polycystic ovarian syndrome. Hum Reprod. 2001 Sep;16(9):1995-8. doi: 10.1093/humrep/16.9.1995. PMID 11527911
- [Background] Parillo F, Zerani M, Maranesi M, Dall'Aglio C, Galeati G, Brecchia G, Boiti C, Gonzalez-Mariscal G. Ovarian hormones and fasting differentially regulate pituitary receptors for estrogen and gonadotropin-releasing hormone in rabbit female. Microsc Res Tech. 2014 Mar;77(3):201-10. doi: 10.1002/jemt.22328. Epub 2013 Dec 26. PMID 24375763
- [Background] Sam S. Obesity and Polycystic Ovary Syndrome. Obes Manag. 2007 Apr;3(2):69-73. doi: 10.1089/obe.2007.0019. No abstract available. PMID 20436797
- [Background] Sir-Petermann T, Codner E, Perez V, Echiburu B, Maliqueo M, Ladron de Guevara A, Preisler J, Crisosto N, Sanchez F, Cassorla F, Bhasin S. Metabolic and reproductive features before and during puberty in daughters of women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2009 Jun;94(6):1923-30. doi: 10.1210/jc.2008-2836. Epub 2009 Feb 17. PMID 19223518
- [Background] Weiner CL, Primeau M, Ehrmann DA. Androgens and mood dysfunction in women: comparison of women with polycystic ovarian syndrome to healthy controls. Psychosom Med. 2004 May-Jun;66(3):356-62. doi: 10.1097/01.psy.0000127871.46309.fe. PMID 15184695